CLINICAL TRIAL: NCT00710515
Title: A Phase I, Open-Label Study to Assess the Effect of Dosing AZD6244 HydSulfate in the Presence and Absence of Food in Patients With Advanced Solid Malignancies
Brief Title: Study to Assess the Effect of Dosing AZD6244 HydSulfate in the Presence and Absence of Food in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1532C00020; 2007-004456-37 EudraCT Number
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Melanoma; Malignant Melanoma
Keywords: Melanoma; Phase I; AZD6244
MeSH Terms: conditions — Melanoma | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): with food
  Interventions: Drug: AZD6244
- 2 (Experimental): without food
  Interventions: Drug: AZD6244

INTERVENTIONS:
Drug: AZD6244 — 75mg

SUMMARY:
The purpose of this study is to test if the levels of AZD6244 in blood are affected by taking food at the same time as the capsules compared to taking capsules on an empty stomach

ELIGIBILITY:
Inclusion Criteria:

* Able to eat a high fat breakfast within a 30-minute period
* Advanced cancer which is refractory to standard therapies, for which no standard therapies exist
* WHO or ECOG performance status 0-2 (those with performance status 2 must have been stable with no deterioration for over 2 weeks)

Exclusion Criteria:

* Any radiotherapy or chemotherapy within 21 days prior to starting the study treatment (not including palliative radiotherapy at focal sites).
* Any evidence of severe or uncontrolled systemic disease (eg., severe hepatic impairment, severe renal impairment, uncontrolled diabetes, acute uncontrolled infection) or current unstable or uncompensated respiratory or cardiac conditions or peripheral vascular disease including diabetic vasculopathy.
* Refractory nausea and vomiting, chronic GI diseases (eg., inflammatory bowel disease) or significant bowel resection that would preclude adequate absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To assess whether food influences the rate and extent of AZD6244 absorption | Day 1 and Day 10

SECONDARY OUTCOMES:
To determine the pharmacokinetics of both AZD6244 and N-desmethyl AZD6244 in the presence and absence of food | Day 1, 2, 3, 8, 9, and 10
To assess the safety and tolerability of AZD6244 in patients with advanced solid malignancies | screening to 30 day post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Chopra, Study Director — AstraZeneca; Jan Schellens, Principal Investigator — Maastricht
Locations (6):
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Maastricht
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, Headington
  - Research Site, London
  - Research Site, Oxford